CLINICAL TRIAL: NCT03329833
Title: Motivational Interviewing and Physical Activity Change in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda Ehrlich-Jones, Assistant Director of Center for Rehabilitation Outcomes Research, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 90IF0093
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Parkinson's; Motivational Interviewing; Exercise; Motivation
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This study examines how a web-based application and/or motivational interviewing impact a participant's exercise routine compared to an educational control group.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants will be aware which group they are assigned to. Study team members who will be providing assessments will be blinded to the condition the participant is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Motivational Interviewing (Experimental): Participants will talk to a coach on the phone who will employ Motivational Interviewing as a coaching style.
  Interventions: Behavioral: Motivational Interviewing
- Web-Based Application (Experimental): Participants will use a Web-Based Application to track their daily physical activity.
  Interventions: Behavioral: Web-based application
- Combination MI and App (Experimental): Participants will have both a coach by phone who will employ Motivational Interviewing as a coaching style and use a Web-Based Application to track their daily physical activity.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Web-based application
- Educational Program (No Intervention): Participants will get to use a website that contains information relevant to patients with Parkinson's Disease.

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational interviewing will consist of weekly phone calls for two months, bi-weekly phone calls for two months, and monthly phone calls for two months.
  Arms: Combination MI and App; Motivational Interviewing
Behavioral: Web-based application — Web-based application participants will be asked to log activity at least on a daily basis.
  Arms: Combination MI and App; Web-Based Application

SUMMARY:
The purpose of this study is to test the efficacy of a 6-month telephone-based motivational interviewing intervention and a web-based application intervention to improve physical activity in participants with Parkinson's Disease.

DETAILED DESCRIPTION:
Participants will be randomized into one of four groups to examine two separate interventions. The groups are: motivational interviewing (a counseling/coaching style), a web-based application for participants to keep track of their physical activity, a combination of the motivational interviewing and the web-based application, and an educational program on various issues related to Parkinson's Disease. The intervention will last 6 months with a follow-up appointment at 9 months. Participants will be asked to come to Galter Pavilion at Northwestern Memorial Hospital or Shirley Ryan AbilityLab a total of five times over the course of the nine months.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* Age 18 or older
* Physician confirmed diagnosis of PD with Hoehn and Yahr stage ≤3
* Ability to ambulate independently (walker is allowed) for distance of 50 feet or 10 minutes at a time
* Does not meet current CDC physical activity guidelines of 150 minutes of moderate to vigorous physical activity per week
* Currently and plans to have a smartphone, tablet, or computer and access to the internet for the next 9 months
* Willing to monitor activity on their smartphone, tablet, or computer via a web-based application during the 9-month program
* Currently uses the internet in a basic capacity

Exclusion Criteria:

* Inability to speak and understand English
* Has a cardiovascular disorder or other health condition that would make exercise unsafe according to their physician
* Patients who are currently receiving physical therapy or received physical therapy one month prior to study enrollment
* Cognitive impairment as defined by inability to provide informed consent and to self-report feelings and behaviors
* Montreal Cognition Scale (MOCA): rating of less than 24, indicative of cognitive dysfunction
* Patients who indicate it is not recommended they participate in increased physical activity as indicated by the Physical Activity Restriction Questionnaire (PAR-Q)
* Patients who are in other studies that monitor fitness or physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Test the efficacy of the Motivational Interviewing (MI) Intervention and the Web-Based Self-Monitoring Application Intervention by monitoring the change in physical activity using data collected from an Actigraph activity monitor. | Assessment will occur at baseline, 3 months, 6 months and 9 months.
  Participants will wear an Actigraph activity monitor for one week every quarter to collect data about physical activity throughout the duration of the study. Time spent doing physical activity will be compared at each assessment for this outcome.
Test the efficacy of the MI Intervention and the Web-Based Self-Monitoring Application Intervention by monitoring the change in physical activity using the Physical Activity Scale for Individuals with Physical Disabilities (PASIPD). | Assessment will occur at baseline, 3 months, 6 months and 9 months.
  PASIPD is a 13-item 7-day physical activity recall questionnaire designed to evaluate physical activity levels in people with physical disabilities by soliciting information about leisure time activities, household activities, and work- related activities.

SECONDARY OUTCOMES:
Test the efficacy of the Motivational Interviewing (MI) intervention and the Web-Based Self-Monitoring Application Intervention for improving balance using the Berg Balance Scale (BBS). | Assessment will occur at baseline, 3 months, 6 months and 9 months.
  The Berg Balance Scale is a 14-item performance measure to assess static balance and fall risk.
Test the efficacy of the Motivational Interviewing (MI) intervention and the Web-Based Self-Monitoring Application Intervention for improving balance using the Activities-Specific Balance Confidence Scale (ABC). | Assessment will occur at baseline, 3 months, 6 months and 9 months.
  Activities-Specific Balance Confidence Scale is a 16-item self-report measure of confidence in performing various activities of daily living without falling.
Test the efficacy of the Motivational Interviewing (MI) intervention and the Web-Based Self-Monitoring Application Intervention for improving balance using the Unified Parkinson's Disease Rating Scale (UPDRS). | Assessment will occur at baseline, 3 months, 6 months and 9 months.
  The UPDRS is an assessment that monitors the progression of Parkinson's Disease. For this outcome, the "postural stability" portion of the assessment will be used to determine balance improvements.
Test the efficacy of the Motivational Interviewing (MI) intervention and the Web-Based Self-Monitoring Application Intervention for improving quality of life using the assessment measure Neuro-QOL. | Assessment will occur at baseline, 3 months, 6 months and 9 months.
  The Neuro-QOL is a set of self-report measures that assess the health-related quality of life of adults and children with neurological disorders.
Test the efficacy of the Motivational Interviewing (MI) intervention and the Web-Based Self-Monitoring Application Intervention for improving quality of life using the assessment measure Patient-Reported Outcomes Measurement Information System (PROMIS). | Assessment will occur at baseline, 3 months, 6 months and 9 months.
  PROMIS Global Health is a 10-item scale rating physical and mental health and overall quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ehrlich-Jones, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (2):
- United States (2):
  - Northwestern Medicine, Chicago, Illinois
  - Shirley Ryan Abilitylab, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stuart M, Chard S, Benvenuti F, Steinwachs S. Community exercise: a vital component to healthy aging. Healthc Pap. 2009;10(1):23-8; discussion 79-83. doi: 10.12927/hcpap.2009.21219. PMID 20057213
- [Background] Brown DR, Yore MM, Ham SA, Macera CA. Physical activity among adults >or=50 yr with and without disabilities, BRFSS 2001. Med Sci Sports Exerc. 2005 Apr;37(4):620-9. doi: 10.1249/01.mss.0000158189.17546.ed. PMID 15809561
- [Background] Ahlskog JE. Does vigorous exercise have a neuroprotective effect in Parkinson disease? Neurology. 2011 Jul 19;77(3):288-94. doi: 10.1212/WNL.0b013e318225ab66. PMID 21768599
- [Background] Alberts JL, Linder SM, Penko AL, Lowe MJ, Phillips M. It is not about the bike, it is about the pedaling: forced exercise and Parkinson's disease. Exerc Sport Sci Rev. 2011 Oct;39(4):177-86. doi: 10.1097/JES.0b013e31822cc71a. PMID 21799425
- [Background] Angevaren M, Aufdemkampe G, Verhaar HJ, Aleman A, Vanhees L. Physical activity and enhanced fitness to improve cognitive function in older people without known cognitive impairment. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005381. doi: 10.1002/14651858.CD005381.pub3. PMID 18646126
- [Background] Bezard E, Yue Z, Kirik D, Spillantini MG. Animal models of Parkinson's disease: limits and relevance to neuroprotection studies. Mov Disord. 2013 Jan;28(1):61-70. doi: 10.1002/mds.25108. Epub 2012 Jul 2. PMID 22753348
- [Background] Chen H, Zhang SM, Schwarzschild MA, Hernan MA, Ascherio A. Physical activity and the risk of Parkinson disease. Neurology. 2005 Feb 22;64(4):664-9. doi: 10.1212/01.WNL.0000151960.28687.93. PMID 15728289
- [Background] Cruise KE, Bucks RS, Loftus AM, Newton RU, Pegoraro R, Thomas MG. Exercise and Parkinson's: benefits for cognition and quality of life. Acta Neurol Scand. 2011 Jan;123(1):13-9. doi: 10.1111/j.1600-0404.2010.01338.x. PMID 20199518
- [Background] van Nimwegen M, Speelman AD, Hofman-van Rossum EJ, Overeem S, Deeg DJ, Borm GF, van der Horst MH, Bloem BR, Munneke M. Physical inactivity in Parkinson's disease. J Neurol. 2011 Dec;258(12):2214-21. doi: 10.1007/s00415-011-6097-7. Epub 2011 May 26. PMID 21614433
- [Background] Ellis T, Boudreau JK, DeAngelis TR, Brown LE, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Dibble LE. Barriers to exercise in people with Parkinson disease. Phys Ther. 2013 May;93(5):628-36. doi: 10.2522/ptj.20120279. Epub 2013 Jan 3. PMID 23288910
- [Background] Ravesloot C. Changing stage of readiness for physical activity in Medicaid beneficiaries with physical impairments. Health Promot Pract. 2009 Jan;10(1):49-57. doi: 10.1177/1524839906292182. Epub 2008 Mar 4. PMID 18319446
- [Background] Harland J, White M, Drinkwater C, Chinn D, Farr L, Howel D. The Newcastle exercise project: a randomised controlled trial of methods to promote physical activity in primary care. BMJ. 1999 Sep 25;319(7213):828-32. doi: 10.1136/bmj.319.7213.828. PMID 10496829
- [Background] Ehrlich-Jones L, Mallinson T, Fischer H, Bateman J, Semanik PA, Spring B, Ruderman E, Chang RW. Increasing physical activity in patients with arthritis: a tailored health promotion program. Chronic Illn. 2010 Dec;6(4):272-81. doi: 10.1177/1742395309351243. Epub 2010 Aug 9. PMID 20696695
- [Background] Brodie DA, Inoue A, Shaw DG. Motivational interviewing to change quality of life for people with chronic heart failure: a randomised controlled trial. Int J Nurs Stud. 2008 Apr;45(4):489-500. doi: 10.1016/j.ijnurstu.2006.11.009. Epub 2007 Jan 26. PMID 17258218
- [Background] Tse MM, Vong SK, Tang SK. Motivational interviewing and exercise programme for community-dwelling older persons with chronic pain: a randomised controlled study. J Clin Nurs. 2013 Jul;22(13-14):1843-56. doi: 10.1111/j.1365-2702.2012.04317.x. Epub 2013 Jan 2. PMID 23279630
- [Background] Haapala I, Barengo NC, Biggs S, Surakka L, Manninen P. Weight loss by mobile phone: a 1-year effectiveness study. Public Health Nutr. 2009 Dec;12(12):2382-91. doi: 10.1017/S1368980009005230. Epub 2009 Mar 27. PMID 19323865
- [Background] Kirwan M, Duncan MJ, Vandelanotte C, Mummery WK. Using smartphone technology to monitor physical activity in the 10,000 Steps program: a matched case-control trial. J Med Internet Res. 2012 Apr 20;14(2):e55. doi: 10.2196/jmir.1950. PMID 22522112
- [Background] Stephens J, Allen J. Mobile phone interventions to increase physical activity and reduce weight: a systematic review. J Cardiovasc Nurs. 2013 Jul-Aug;28(4):320-9. doi: 10.1097/JCN.0b013e318250a3e7. PMID 22635061
- [Background] Olanow CW, Stern MB, Sethi K. The scientific and clinical basis for the treatment of Parkinson disease (2009). Neurology. 2009 May 26;72(21 Suppl 4):S1-136. doi: 10.1212/WNL.0b013e3181a1d44c. PMID 19470958
- [Background] O'Brien J, Ward A, Michels S, Tzivelekis S, Brandt N. Economic burden associated with Parkinson disease. Drug Benefit Trends. 2009;21(6):179-190.
- [Background] Chen JJ. Parkinson's disease: health-related quality of life, economic cost, and implications of early treatment. Am J Manag Care. 2010 Mar;16 Suppl Implications:S87-93. PMID 20297871
- [Background] Shulman LM, Gruber-Baldini AL, Anderson KE, Vaughan CG, Reich SG, Fishman PS, Weiner WJ. The evolution of disability in Parkinson disease. Mov Disord. 2008 Apr 30;23(6):790-6. doi: 10.1002/mds.21879. PMID 18361474
- [Background] Goodwin VA, Richards SH, Taylor RS, Taylor AH, Campbell JL. The effectiveness of exercise interventions for people with Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2008 Apr 15;23(5):631-40. doi: 10.1002/mds.21922. PMID 18181210
- [Background] Ashburn A, Fazakarley L, Ballinger C, Pickering R, McLellan LD, Fitton C. A randomised controlled trial of a home based exercise programme to reduce the risk of falling among people with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):678-84. doi: 10.1136/jnnp.2006.099333. Epub 2006 Nov 21. PMID 17119004
- [Background] Ellis T, Motl RW. Physical activity behavior change in persons with neurologic disorders: overview and examples from Parkinson disease and multiple sclerosis. J Neurol Phys Ther. 2013 Jun;37(2):85-90. doi: 10.1097/NPT.0b013e31829157c0. PMID 23632452
- [Background] van Nimwegen M, Speelman AD, Smulders K, Overeem S, Borm GF, Backx FJ, Bloem BR, Munneke M; ParkFit Study Group. Design and baseline characteristics of the ParkFit study, a randomized controlled trial evaluating the effectiveness of a multifaceted behavioral program to increase physical activity in Parkinson patients. BMC Neurol. 2010 Aug 19;10:70. doi: 10.1186/1471-2377-10-70. PMID 20723221
- [Background] Fazio P, Granieri G, Casetta I, Cesnik E, Mazzacane S, Caliandro P, Pedrielli F, Granieri E. Gait measures with a triaxial accelerometer among patients with neurological impairment. Neurol Sci. 2013 Apr;34(4):435-40. doi: 10.1007/s10072-012-1017-x. Epub 2012 Mar 25. PMID 22447360
- [Background] Dijkstra B, Zijlstra W, Scherder E, Kamsma Y. Detection of walking periods and number of steps in older adults and patients with Parkinson's disease: accuracy of a pedometer and an accelerometry-based method. Age Ageing. 2008 Jul;37(4):436-41. doi: 10.1093/ageing/afn097. Epub 2008 May 16. PMID 18487266
- [Background] Strath SJ, Kaminsky LA, Ainsworth BE, Ekelund U, Freedson PS, Gary RA, Richardson CR, Smith DT, Swartz AM; American Heart Association Physical Activity Committee of the Council on Lifestyle and Cardiometabolic Health and Cardiovascular, Exercise, Cardiac Rehabilitation and Prevention Committee of the Council on Clinical Cardiology, and Council. Guide to the assessment of physical activity: Clinical and research applications: a scientific statement from the American Heart Association. Circulation. 2013 Nov 12;128(20):2259-79. doi: 10.1161/01.cir.0000435708.67487.da. Epub 2013 Oct 14. PMID 24126387
- [Background] Ham SA, Reis JP, Strath SJ, Dubose KD, Ainsworth BE. Discrepancies between methods of identifying objectively determined physical activity. Med Sci Sports Exerc. 2007 Jan;39(1):52-8. doi: 10.1249/01.mss.0000235886.17229.42. PMID 17218884
- [Background] Martins RK, McNeil DW. Review of Motivational Interviewing in promoting health behaviors. Clin Psychol Rev. 2009 Jun;29(4):283-93. doi: 10.1016/j.cpr.2009.02.001. Epub 2009 Feb 23. PMID 19328605
- [Background] Rochester L, Chastin SF, Lord S, Baker K, Burn DJ. Understanding the impact of deep brain stimulation on ambulatory activity in advanced Parkinson's disease. J Neurol. 2012 Jun;259(6):1081-6. doi: 10.1007/s00415-011-6301-9. Epub 2011 Nov 16. PMID 22086738
- [Background] Smith DC, Lanesskog D, Cleeland L, Motl R, Weikert M, Dlugonski D. Motivational interviewing may improve exercise experience for people with multiple sclerosis: A small randomized trial. Health Soc Work. 2012 May;37(2):99-109. doi: 10.1093/hsw/hls011. PMID 23029977
- [Background] Wallen MB, Dohrn IM, Stahle A, Franzen E, Hagstromer M. Comparison of pedometer and accelerometer derived steps in older individuals with Parkinson's disease or osteoporosis under free-living conditions. J Aging Phys Act. 2014 Oct;22(4):550-6. doi: 10.1123/japa.2013-0052. Epub 2013 Dec 4. PMID 24306767
- [Background] Washburn RA, Zhu W, McAuley E, Frogley M, Figoni SF. The physical activity scale for individuals with physical disabilities: development and evaluation. Arch Phys Med Rehabil. 2002 Feb;83(2):193-200. doi: 10.1053/apmr.2002.27467. PMID 11833022
- [Background] van den Berg-Emons RJ, L'Ortye AA, Buffart LM, Nieuwenhuijsen C, Nooijen CF, Bergen MP, Stam HJ, Bussmann JB. Validation of the Physical Activity Scale for individuals with physical disabilities. Arch Phys Med Rehabil. 2011 Jun;92(6):923-8. doi: 10.1016/j.apmr.2010.12.006. Epub 2011 Apr 19. PMID 21507382
- [Background] Lun V, Pullan N, Labelle N, Adams C, Suchowersky O. Comparison of the effects of a self-supervised home exercise program with a physiotherapist-supervised exercise program on the motor symptoms of Parkinson's disease. Mov Disord. 2005 Aug;20(8):971-5. doi: 10.1002/mds.20475. PMID 15838853
- [Background] Qutubuddin AA, Pegg PO, Cifu DX, Brown R, McNamee S, Carne W. Validating the Berg Balance Scale for patients with Parkinson's disease: a key to rehabilitation evaluation. Arch Phys Med Rehabil. 2005 Apr;86(4):789-92. doi: 10.1016/j.apmr.2004.11.005. PMID 15827933
- [Background] Conradsson D, Lofgren N, Stahle A, Hagstromer M, Franzen E. A novel conceptual framework for balance training in Parkinson's disease-study protocol for a randomised controlled trial. BMC Neurol. 2012 Sep 27;12:111. doi: 10.1186/1471-2377-12-111. PMID 23017069
- [Background] Mhatre PV, Vilares I, Stibb SM, Albert MV, Pickering L, Marciniak CM, Kording K, Toledo S. Wii Fit balance board playing improves balance and gait in Parkinson disease. PM R. 2013 Sep;5(9):769-77. doi: 10.1016/j.pmrj.2013.05.019. Epub 2013 Jun 11. PMID 23770422
- [Background] Lim LI, van Wegen EE, de Goede CJ, Jones D, Rochester L, Hetherington V, Nieuwboer A, Willems AM, Kwakkel G. Measuring gait and gait-related activities in Parkinson's patients own home environment: a reliability, responsiveness and feasibility study. Parkinsonism Relat Disord. 2005 Jan;11(1):19-24. doi: 10.1016/j.parkreldis.2004.06.003. PMID 15619458
- [Background] Hesse BW, Hanna C, Massett HA, Hesse NK. Outside the box: will information technology be a viable intervention to improve the quality of cancer care? J Natl Cancer Inst Monogr. 2010;2010(40):81-9. doi: 10.1093/jncimonographs/lgq004. PMID 20386056
- [Background] Abras C, Maloney-Krichmar D, Preece J. User-centered design. In: Bainbridge W, ed. Berkshire Encyclopedia of Human-Computer Interaction. Great Barrington, MA: Berkshire Publishing Group; 2004:463-468
- [Background] Brinck T, Gergle D, Wood S. Usability for the Web: Designing Web Sites that Work. San Francisco, CA: Morgan Kaufmann Publishers; 2002.
- [Background] Nielsen J, Loranger H. Prioritizing web usability. Berkley, CA: New Riders Press; 2006.
- [Background] Badke MB, Shea TA, Miedaner JA, Grove CR. Outcomes after rehabilitation for adults with balance dysfunction. Arch Phys Med Rehabil. 2004 Feb;85(2):227-33. doi: 10.1016/j.apmr.2003.06.006. PMID 14966706
- [Background] Hebert JS, Wolfe DL, Miller WC, Deathe AB, Devlin M, Pallaveshi L. Outcome measures in amputation rehabilitation: ICF body functions. Disabil Rehabil. 2009;31(19):1541-54. doi: 10.1080/09638280802639467. PMID 19479495
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984